CLINICAL TRIAL: NCT02260063
Title: A Trial in Healthy Volunteers of the Relative Bioavailability of Epinastine Syrup, a New Galenic Form, Compared to the Reference Product Tablets
Brief Title: Relative Bioavailability of Epinastine Syrup Compared to Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 262.252
Record Dates: First submitted 2014-10-08; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — epinastine

ARMS (2):
- Epinastine syrup (Experimental)
  Interventions: Drug: Epinastine syrup
- Epinastine tablets (Active Comparator)
  Interventions: Drug: Epinastine tablets

INTERVENTIONS:
Drug: Epinastine syrup
  Arms: Epinastine syrup
Drug: Epinastine tablets
  Arms: Epinastine tablets

SUMMARY:
To assess the bioequivalence of two galenic formulations for epinastine (Flurinol®): syrup and 20 mg tablets

ELIGIBILITY:
Inclusion Criteria:

* male and female, non-smoker and non-alcohol user, healthy volunteers, of 21 - 45 years of age. To be eligible, women must not be pregnant or lactating and they must not be taking hormone contraceptives
* Volunteers must not have a history of liver or renal disease or a history of psychiatric disorder. Volunteers will be submitted to the biochemical tests listed below, the results of which must be within expected normal values: complete blood count, erythro-sedimentation rate, GOT (glutamate oxalacetate transaminase) GPT (glutamate pyruvate transaminase), blood creatinine, glycemia, uremia, blood cholesterol, pregnancy test. HIV test (with prior written consent), serum tests for Chagas disease, hepatic b and syphilis, complete urinalysis, ECG (electrocardiogram) and chest x-ray
* Volunteers must have discontinued all pharmacological treatment at least two weeks before entering this trial
* informed written consent, signed prior to the start of this trial

Exclusion Criteria:

* Volunteers requiring any kind of pharmacological treatment or having some known addiction
* Volunteers having participated in any other clinical trial during the four preceding weeks
* Volunteers who must start a treatment incompatible with this trial during its course
* Volunteers who do not comply with the fasting requirements established in the trial or who do not comply with trial requirements such as avoiding intake of coffee, tea, cola soft drinks, etc. for 24 hours prior to the start of the trial
* History of allergy or intolerance to Epinastine
* Uncooperative volunteers
* Previous participation in this trial

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 1998-11; Primary Completion 1999-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of plasma concentration (CP) | Up to 24 hours after drug administration
Absorption rate Cpmax/AUC | Up to 24 hours after drug administration

SECONDARY OUTCOMES:
Peak plasma concentration (Cpmax) | Up to 24 hours after drug administration
Time to peak (Tmax) | Up to 24 hours after drug administration
Drug half - life (T1/2) | Up to 24 hours after drug administration
Number of participants with adverse events | Up to 24 hours after last drug administration
Number of participants withdrawn or discontinued due to safety reasons | Up to 24 hours after last drug administration
Number of participants with abnormal findings in physical examination | Up to 24 hours after last drug administration
Number of participants with clinically significant findings in vital signs | Up to 24 hours after last drug administration